CLINICAL TRIAL: NCT01568450
Title: A Randomized, Open-label, Single-dose, Crossover Study to Investigate The Pharmacokinetics Between a GL2907 XL and Oxycontin CR Tab. 10mg in Healthy Male Volunteers
Brief Title: A Open-label, Single-dose Study to Investigate The Pharmacokinetics Between a GL2907 XL and Oxycontin CR Tab. 10mg in Healthy Male Volunteers
Acronym: GL2907-101
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GL Pharm Tech Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: GL2907-101
Record Dates: First submitted 2012-03-19; First posted 2012-04-02 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2013-01

CONDITIONS: Healthy
Keywords: Oxycodone, controlled release formulation
MeSH Terms: interventions — Oxycodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- GL2907 XL 20mg (Oxycodone 20mg, fasted) (Experimental)
  Interventions: Drug: Oxycodone
- GL2907 XL 20mg (Oxycodone 20mg, after high fat meal) (Experimental)
  Interventions: Drug: Oxycodone
- Oxycontin CR 10mg (Oxycodone 10mg, fasted) (Active Comparator)
  Interventions: Drug: Oxycodone

INTERVENTIONS:
Drug: Oxycodone — Oxycodone XL 20mg(20mg once a day, fasted)
  Arms: GL2907 XL 20mg (Oxycodone 20mg, fasted)
Drug: Oxycodone — Oxycodone XL 20mg/day(20mg once a day, after high fat meal)
  Arms: GL2907 XL 20mg (Oxycodone 20mg, after high fat meal)
Drug: Oxycodone — Oxycodone 20mg/day (10mg twice a day, fasted)
  Arms: Oxycontin CR 10mg (Oxycodone 10mg, fasted)

SUMMARY:
The purpose of this clinical trial is to compare the pharmacokinetic characteristics of GL2907 XL 20mg tablet and Oxycontin CR 10mg tablet.

GL2907 XL 20mg tablet is controlled released formulation which is made by GL Pharm Tech.

ELIGIBILITY:
Inclusion Criteria:

* 20~45 years old, Healthy Adult Male Subject
* ≥ 50kg(Body Weight) and Ideal Body Weight ≤ ±20%

Exclusion Criteria:

* ALT or AST > 1.25(Upper Normal Range)
* Total Bilirubin > 1.5 (Upper Normal Range)
* BUN or Creatinine > Normal Range
* Systolic BP > 160mmHg or < 80mmHg, Diastolic BP > 100mmHg or < 50mmHg

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-03; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Cmax | 48hr
  Pharmacokinetic of Oxycodone
AUC(0-24h) | 24 hr
  Pharmacokinetic of Oxycodone

SECONDARY OUTCOMES:
Tmax | 48 hr
  Pharmacokinetic of Oxycodone
t1/2 | 48 hr
  Pharmacokinetic of Oxycodone
Vz/F | 48 hr
  Pharmacokinetic of Oxycodone
CL/F | 48 hr
  Pharmacokinetic of Oxycodone
Safety Monitoring | 27 days
  Adverse Event, Vital sign, 12-lead ECG, Physical Exam, Laboratory test

CONTACTS AND LOCATIONS:
Overall Officials: Doo-Yeoun Cho, MD, Principal Investigator — Ajou University School of Medicine
Locations (1):
- AJOU University Hospital, Suwon, Gyeonggido, South Korea